CLINICAL TRIAL: NCT02583763
Title: Cardiac Displacement From Third Trimester to Early Childhood
Acronym: CADETTE
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Ostergotland County Council, Sweden (Other); Stiftelsen Samariten (Other)
Responsible Party: Principal Investigator, Olov Änghagen, Paediatrician, PhD student, University Hospital, Linkoeping
Other Study IDs: 2012/257-31
Record Dates: First submitted 2015-10-16; First posted 2015-10-22 (Estimated); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: IUGR; Fetal Growth Retardation; Intrauterine Growth Restriction
Keywords: pro-brain natriuretic peptide (1-76); Insulin-Like Growth Factor Binding Proteins; Insulin-Like Growth Factor I; Echocardiography; Velocity Vector Imaging; Heart Function Tests
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Years
Biospecimen Retention: Samples With DNA — The investigators will take a blood sample from the umbilical cord at birth and again at 9 years of age. The sample will be analyzed for growth factors and cardiac markers.
  2015-05-20 an additional ethical approval was accepted for analyzing epigenetic factors in the children's DNA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fetuses/Children with IUGR: The moving sequences of the heart movement are collected at the regular ultrasound examinations during pregnancy. Following delivery the investigators plan to examine the baby with cardiac ultrasound, echocardiography, between 12 and 72 hours after delivery and again when the child is 3-4 months old and at 9 years of age.
  Blood sample will be taken from the umbilical cord at birth and again at 9 years of age. The investigators will analyse the blood for growth factors and cardiac markers. An additional ethical approval was accepted 2015 for analysing epigenetic factors in the children's DNA.
  Due to corona pandemic the follow up was delayed from 7 to 9 years of age. Approved by the ethical committee.
  Interventions: Other: Echocardiography; Procedure: Blood sample
- Healthy Controls: The moving sequences of the heart movement are collected at two occasions approximately 4 weeks apart. This takes place during gestational weeks 28-36. Following delivery the investigators plan to examine the baby with cardiac ultrasound, echocardiography, between 12 and 72 hours after delivery and again when the child is 3-4 months old and at 9 years of age.
  Blood sample will be taken from the umbilical cord at birth and again at 9 years of age. The investigators will analyze the blood for growth factors and cardiac markers. An additional ethical approval was accepted 2015 for analysing epigenetic factors in the children's DNA.
  Due to corona pandemic the follow up was delayed from 7 to 9 years of age. Approved by the ethical committee.
  Interventions: Other: Echocardiography; Procedure: Blood sample

INTERVENTIONS:
Other: Echocardiography — During the ultrasound examinations standardized, moving sequences of the heart will be saved. Analyzes are performed off-line and analyzed by vector velocity imaging software.
Procedure: Blood sample — The investigators will take a blood sample from the umbilical cord at birth and again at 9 years of age.

SUMMARY:
The aim is to increase awareness of the relationship between (IUGR) and cardiac function in the foetus, the development of cardiac function over time after delivery and what significance a possible early disturbed myocardial function have for the neonate and the child during the first years of life.

DETAILED DESCRIPTION:
This is a prospective case-control study in which fetuses from normal pregnancies will be compared with fetuses with IUGR. Parents will be asked to participate in the study in connection with the routine ultrasound examinations at the department of obstetrics to where they have been referred because of suspected IUGR. The control group will be randomly selected among pregnant women who come for routine ultrasound during pregnancy at gestational week 18-20.

Surveys will be performed in the third trimester and after delivery. During the ultrasound examinations standardized, moving sequences of the heart will be saved. Analyses will be performed off-line and analysed by vector velocity imaging software. With this technique, the investigator can quantify the chamber wall and myocardial movements. Speed (velocity), movement (displacement) and thickening/deformation (strain and strain rate) will be recorded in a structured and standardized manner.

When performing the analysis the heart's walls are outlined and the software extracts the movement in different directions.

Data will be obtained concerning the participating mothers previous illness, mothers' age, maternal smoking, BMI, any abnormalities during pregnancy, number of previous pregnancies. Other data that will be recorded are means of delivery and any abnormalities during previous pregnancies, such as hypertension, preeclampsia and pre-natal steroid treatment.

Additional data to be collected from the participating fetuses are flow profiles in the umbilical artery, ductus venosus and middle cerebral artery. Abdominal circumference and estimated weight will be registered.

Following delivery, the participating child's height, weight, head circumference and gestational age at birth are registered. Additional data that will be collected after delivery are umbilical vein and umbilical artery acid base values, Apgar score. If admitted to the pediatric ward the investigators will register the number of days hospitalized in the ward for post-natal care and diagnosis. The investigators plan to examine the participating baby with cardiac ultrasound between 12 and 72 hours after delivery and again when the participating child is 3-4 months old and at 7-9 years of age.

The investigators will take a blood sample from the umbilical cord at birth and again at 7-9 years of age. The investigators will analyse the blood for growth factors and cardiac markers. An additional ethical approval was accepted 2015 for analysing epigenetic factors in the participating children's DNA.

Based on power calculation the investigators plan to examine between 20-30 fetuses with IUGR and 40-60 healthy fetuses in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion of research subjects: Growth restriction in routine pregnancy ultrasound, verified by specialist control. Gestational age based on Crown Rump Length measurements during the first trimester. Growth restriction defined by a deviation more than 22% from the normal curve at a given gestational age or growth rate deviates more than 10% compared to the previous measurement in relation to the expected weight.
* Inclusion of controls: Control individuals recruited among mothers who come to routine pregnancy ultrasound control at gestational week 18. These are randomly selected and then asked to participate.

Exclusion Criteria:

* Exclusion of both the cases with IUGR and the control cases are major malformations, twin pregnancy, signs of intrauterine infection during pregnancy, significant illness or significant medical treatment of the mother.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is a prospective case-control study in which fetuses from normal pregnancies will be compared with fetuses with IUGR. Parents will be asked to participate in the study in connection with the routine ultrasound examinations at the department of obstetrics to where they have been referred because of suspected IUGR. The control group will be randomly selected among pregnant women who come for routine ultrasound during pregnancy at gestational week 18-20.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2027-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Olov Änghagen, PhD student, Principal Investigator — Dept of Paediatric, Linköping; Nina Nelson, Professor, Study Chair — Karolinska University Hospital, Stockholm; Peter Bang, Professor, Study Chair — Dept of Paediatric, Linköping; Jan Engvall, Professor, Study Chair — Dept of Clinical Physiology, Linköping; Eva Nylander, Professor, Study Chair — Dept of Clinical Physiology, Linköping
Locations (2):
- Sweden (2):
  - Dept of Obstetrics and Gynecology, Linköping
  - Paediatric Department University Hospital, Linköping

REFERENCES:
- [Derived] Anghagen O, Engvall J, Gottvall T, Nelson N, Nylander E, Bang P. Developmental Differences in Left Ventricular Strain in IUGR vs. Control Children the First Three Months of Life. Pediatr Cardiol. 2022 Aug;43(6):1286-1297. doi: 10.1007/s00246-022-02850-y. Epub 2022 Mar 25. PMID 35333947

RESULTS

PARTICIPANT FLOW:
Groups:
- Fetuses/Children With IUGR: The moving sequences of the heart movement are collected at the regular ultrasound examinations during pregnancy. Following delivery the investigators plan to examine the baby with cardiac ultrasound, echocardiography, between 12 and 72 hours after delivery and again when the child is 3-4 months old and at 7 years of age.
  Blood sample will be taken from the umbilical cord at birth and again at 7 years of age. The investigators will analyse the blood for growth factors and cardiac markers. An additional ethical approval was accepted 2015 for analysing epigenetic factors in the children's DNA.
  Echocardiography: During the ultrasound examinations standardized, moving sequences of the heart will be saved. Analyzes are performed off-line and analyzed by vector velocity imaging software.
  Blood sample: The investigators will take a blood sample from the umbilical cord at birth and again at 7 years of age.
- Healthy Controls: The moving sequences of the heart movement are collected at two occasions approximately 4 weeks apart. This takes place during gestational weeks 28-36. Following delivery the investigators plan to examine the baby with cardiac ultrasound, echocardiography, between 12 and 72 hours after delivery and again when the child is 3-4 months old and at 7 years of age.
  Blood sample will be taken from the umbilical cord at birth and again at 7 years of age. The investigators will analyze the blood for growth factors and cardiac markers. An additional ethical approval was accepted 2015 for analysing epigenetic factors in the children's DNA.
  Echocardiography: During the ultrasound examinations standardized, moving sequences of the heart will be saved. Analyzes are performed off-line and analyzed by vector velocity imaging software.
  Blood sample: The investigators will take a blood sample from the umbilical cord at birth and again at 7 years of age.
Period: Overall Study
Arm/Group | Fetuses/Children With IUGR | Healthy Controls
Started | 21 | 40
Completed | 18 | 35
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fetuses/Children With IUGR | Healthy Controls | Total
Number analyzed (Participants) | 18 | 35 | 53
Age, Continuous [Mean (Standard Deviation); unit: Gestational age] | 36.4 (3.9) | 39.7 (1.5) | 36.6 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 17 | 25
  Male | 10 | 18 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Velocity of the Cardiac Walls cm/s Divided With Chamber Length in mm = Quota cm/s / mm
Description: Echocardiography images of the heart's walls are outlined and the software extracts the movement in different directions. At each timepoint offline calculation were performed three times on each image and an averaged was calculated.
  The length of the heart from the level of the AV valve to the apex in left ventricle is used as a measurement for the size of the heart.
  As the velocity increases when the size of the heart increases a quota is used dividing the velocity by the length of the heart to be able to compare the velocity at different timepoints whe the child is growing.
  Quota=Left chamber velocity at septum stated in cm/s divided by ventricular length in mm.
Time Frame: After delivery echocardiography were performed. This is one time point. Due to the known dramatic hemodynamic changes for all children right after birth we defined this time point to somewhere between 12 and 72 hours of age.
Measure: Mean (Standard Deviation); unit: cm/s/mm = quota
Groups:
- Fetuses/Children With Fetal Growth Restriction: Growth restriction was defined as a prenatal estimated weight deviation more than 22% from the normal curve at a given gestational age or growth rate deviating more than 10% compared to the previous measurement in relation to the expected weight.
- Healthy Controls: Fetuses in a control group were randomly selected among pregnant women who came for routine ultrasound during pregnancy at gestational week 18-20 having normal fetal examination with a normal estimated birth weight.
Arm/Group | Fetuses/Children With Fetal Growth Restriction | Healthy Controls
Number analyzed (Participants) | 18 | 35
cm/s/mm = quota | 0,095 (0,018) | 0,087 (0,016)
Statistical Analysis 1: Comparison: Fetuses/Children With Fetal Growth Restriction vs Healthy Controls; Paired sample T test were used to analyse normally distributed data; Test type: Superiority; p > 0.05, t-test, 2 sided — Significance value stated as p<0.05

2. Secondary Outcome: Left Chamber Longitudinal Displacement in the Septal Wall at the AV Valve Level Corrected for Ventricular Length Expressed as a Ratio.
Description: Echocardiography images of the heart's walls are outlined and the software extracts the movement in mm in the myocardial wall from end diastole to end systole.
  The movement of the myocardium from end diastole to end systole at the AV valve level of the septal wall is measured in mm and expressed as a ratio compared to the ventricular length in mm at the end of diastole.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/mm = ratio
Groups:
- Fetuses/Children With Fetal Growth Restriction: Growth restriction was defined as a deviation more than 22% from the normal curve at a given gestational age or growth rate deviating more than 10% compared to the previous measurement in relation to the expected weight.
- Healthy Controls: The moving sequences of the heart movement are collected at two occasions approximately 4 weeks apart. This takes place during gestational weeks 28-36. Following delivery the investigators plan to examine the baby with cardiac ultrasound, echocardiography. First examination is between 12 and 72 hours after delivery and second examination is when the child is 3 months old and at the third examination is at 9 years of age.
  Blood sample will be taken from the umbilical cord at birth and again at 9 years of age. The investigators will analyze the blood for growth factors and cardiac markers. An additional ethical approval was accepted 2015 for analysing epigenetic factors in the children's DNA.
  Due to corona pandemic the follow up was delayed from 7 to 9 years of age. Approved by the ethical committee.
  Echocardiography: During the ultrasound examinations standardized, moving sequences of the heart will be saved. Analyzes are performed off-line and analyzed by vector velocity imaging software.
  Blood sample: The investigators will take a blood sample from the umbilical cord at birth and again at 9 years of age.
Arm/Group | Fetuses/Children With Fetal Growth Restriction | Healthy Controls
Number analyzed (Participants) | 18 | 35
mm/mm = ratio | 0,112 (0,026) | 0,110 (0,028)
Statistical Analysis 1: Comparison: Fetuses/Children With Fetal Growth Restriction vs Healthy Controls; Test type: Superiority; p > 0.05, t-test, 2 sided — Significance value was stated as p<0.05

3. Secondary Outcome: Average Longitudinal 4 Segmental Strain in the Cardiac Wall. Shortening of the Myocardium in Systole.
Description: Echocardiography images of the heart's walls are outlined and the software extracts the movement in different directions.
  A 4 chamber view of the hartt is used and calculation of 6 segments (2 basal, 2 mid and 2 apical segments) were performed three times on each image and an averaged was calculated. The 2 basal segments closeset to the AV valve and the two 2 mid segments were summed and averaged into average longitudinal 4 segmental strain.
  Strain in % is the averege shortening of the myocardium in systole.
Time Frame: At 3 months
Population: Average longitudinal 4 segmental myocardial strain at 3 months of age
Measure: Mean (Standard Deviation); unit: percentage of myocardium shortening.
Groups:
- Fetuses/Children With Fetal Growth Restriction: Growth restriction was defined as a prenatal estimated weightdeviation more than 22% from the normal curve at a given gestational age or growth rate deviating more than 10% compared to the previous measurement in relation to the expected weight.
Arm/Group | Fetuses/Children With Fetal Growth Restriction | Healthy Controls
Number analyzed (Participants) | 18 | 35
percentage of myocardium shortening. | -17.8 (3.82) | -20.92 (3.31)
Statistical Analysis 1: Comparison: Fetuses/Children With Fetal Growth Restriction vs Healthy Controls; Test type: Superiority; p = 0.003, t-test, 2 sided — Significance value was set to p<0.05

4. Secondary Outcome: Cardiac Marker Troponin T
Description: Comparing cardiac marker troponin T between the two groups
Time Frame: At birth and at 9 years of age
Reporting Status: Not Posted, anticipated posting 2028-12

5. Secondary Outcome: Cardiac Marker N-terminal Prohormone of Brain Natriuretic Peptide (NT-ProBNP)
Description: Comparing N-terminal prohormone of brain natriuretic peptide marker NT-ProBNP between the two groups
Time Frame: At birth and at 9 years of age
Reporting Status: Not Posted, anticipated posting 2028-12

6. Secondary Outcome: Insulin-like Growth Factor-1 (IGF-1)
Description: Comparing IGF-1 between the two groups
Time Frame: At birth and at 9 years of age
Reporting Status: Not Posted, anticipated posting 2028-12

7. Secondary Outcome: Insulin-like Growth Factor Binding Protein (IGFBP)
Description: Comparing Insulin-like growth factor binding protein (IGFBP) between the two groups
Time Frame: At birth and at 9years of age
Reporting Status: Not Posted, anticipated posting 2028-12

8. Secondary Outcome: DNA Methylation and Gene Expression in Blood Monocytes and Lymphocytes
Description: Changes in DNA methylation and gene expression will be compared between the two groups
Time Frame: At birth and at 9 years of age
Reporting Status: Not Posted, anticipated posting 2028-12

ADVERSE EVENTS:
Time Frame: Time frame from inclusion to 9 years of age with 3 specific timepoints of follow-ups. at 12-72 hours of age. at 3- 4 months of age at 9 years of age.
Description: As this is an observational study we do not introduce any extra risk for the children when participating in the study
Arm/Group | Fetuses/Children With IUGR | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 2/18 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/35
Other Adverse Events (participants affected / at risk) | 0/18 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2014-03-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT02583763/Prot_000.pdf